CLINICAL TRIAL: NCT04967066
Title: Serum Levels of Adipocytokines in Children With Febrile Seizures: A Cross-Sectional Study at Sohag University Hospital
Brief Title: A Cross-Sectional Study of Serum Levels of Adipocytokines in Children With Febrile Seizures
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hagar Abdelhamid Mohamed, Resident of Pediatrics, Sohag University Hospital, Sohag University
Other Study IDs: Soh-Med-21-07-06
Record Dates: First submitted 2021-07-13; First posted 2021-07-19 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Febrile Seizure
MeSH Terms: conditions — Seizures, Febrile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples With DNA — The serum will be obtained by centrifugation at 3,500 rpm for 5 min at 4 ℃. The serum will be immediately separated and stored at -70 ℃. Serum leptin and adiponectin will be assessed through enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- children with febrile convulsions: * Inclusion criteria
  * Age from 6 months to 6 years.
  * Seizures.
  * Fever (≥38°C).
  * Exclusion criteria
  * Central nervous system infection.
  * Epilepsy.
  * Previous neurological abnormalities.
  * Inborn errors of metabolism.
  * Immunological diseases.
  * Endocrinal diseases (e.g., diabetes mellitus).
  * Obesity.
  * Eating disorders.
  * Gastrointestinal disorders (e.g., diarrhea).
  Interventions: Diagnostic Test: Serum Levels of Adipocytokines
- Febrile children without convulsions: * Inclusion criteria
  * Age from 6 months to 6 years.
  * Fever (≥38°C) due to acute infection.
  * Exclusion criteria
  * Seizures.
  * Central nervous system infection.
  * Previous neurological abnormalities.
  * Inborn errors of metabolism.
  * Immunological diseases.
  * Endocrinal diseases (e.g., diabetes mellitus).
  * Obesity.
  * Eating disorders.
  * Gastrointestinal disorders (e.g., diarrhea).
  Interventions: Diagnostic Test: Serum Levels of Adipocytokines
- Healthy control children: * Inclusion criteria
  * Age from 6 months to 6 years.
  * Presented for routine check-up.
  * Exclusion criteria
  * Fever.
  * Seizures.
  * Central nervous system infection.
  * Previous neurological abnormalities.
  * Inborn errors of metabolism.
  * Immunological diseases.
  * Endocrinal diseases (e.g., diabetes mellitus).
  * Obesity.
  * Eating disorders.
  * Gastrointestinal disorders (e.g., diarrhea).
  * Any illness in the last month.
  Interventions: Diagnostic Test: Serum Levels of Adipocytokines

INTERVENTIONS:
Diagnostic Test: Serum Levels of Adipocytokines — Serum leptin and adiponectin: venous blood samples (3 ml) will be obtained from children with FS (within 3 hours of seizures) as well as the two control groups. The serum will be obtained by centrifugation at 3,500 rpm for 5 min at 4 ℃. The serum will be immediately separated and stored at -70 ℃. Serum leptin and adiponectin will be assessed through enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions.

SUMMARY:
Febrile seizure (FS) is a common neurological condition in children, affecting 2 - 14% of children. FS is defined as seizures occurring in a child aged from six months to five years that is accompanied by a fever (≥38°C) without central nervous system infection. FS is classified into simple febrile seizure (SFS) and complex febrile seizure (CFS). SFS accounts for 70-75% of FS cases and is characterized by being generalized, duration of less than 15 minutes, occurs once in 24 hours, and no previous neurologic problems. We aim to investigate serum levels of adipocytokines, specifically leptin, adiponectin, and IL-6, in children with FS.

DETAILED DESCRIPTION:
The study will include three groups of children (100 for each): children with febrile seizures (group 1), febrile children without seizures (group 2), and healthy control children (group 3). Children included in this study will undergo:

* Thorough medical history taking: including age, gender, and seizure details for children with febrile seizures (e.g., type, duration, recurrence).
* Physical examination: including vital signs (particularly temperature) and comprehensive neurological examination).
* Laboratory investigations:

  * Routine investigations: complete blood count, C-reactive protein, blood glucose, serum electrolytes (sodium, potassium, calcium, and magnesium), liver and kidney function tests.
  * Serum leptin and adiponectin: venous blood samples (3 ml) will be obtained from children with FS (within 3 hours of seizures) as well as the two control groups. Serum will be obtained by centrifugation at 3,500 rpm for 5 min at 4 ℃. The serum will be immediately separated and stored at -70 ℃. Serum leptin and adiponectin will be assessed through enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* Age from 6 months to 6 years.
* Seizures.
* Fever (≥38°C) due to acute infection.
* Presented for routine check-up.

Exclusion Criteria:

* Central nervous system infection.
* Epilepsy.
* Previous neurological abnormalities.
* Inborn errors of metabolism.
* Immunological diseases.
* Endocrinal diseases (e.g., diabetes mellitus).
* Obesity.
* Eating disorders.
* Gastrointestinal disorders (e.g., diarrhea).
* Seizures.
* Previous neurological abnormalities
* Any illness in the last month

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Chi-square test will be used in comparing qualitative data between two groups, and Fisher exact test will be used instead of the Chi-square test when the expected count in any cell is less than 5. Student's T-test will be used in the comparison between two groups with quantitative data and parametric distribution, and Mann-Whitney test will be used in the comparison between two groups with quantitative data and non-parametric distribution. One-way analysis of variance (ANOVA) and Kruskal-Wallis tests will be used to compare more than two independent groups for quantitative data with parametric and non-parametric distribution, respectively. Pearson's and Spearman's correlation will be used to test the correlation analysis.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Serum leptin | within 3 hours of seizures
  venous blood samples (3 ml) will be obtained from children with FS as well as the two control groups. Serum will be obtained by centrifugation at 3,500 rpm for 5 min at 4 ℃. The serum will be immediately separated and stored at -70 ℃. Serum leptin will be assessed through enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions.
Serum adiponectin | within 3 hours of seizures
  venous blood samples (3 ml) will be obtained from children with FS as well as the two control groups. Serum will be obtained by centrifugation at 3,500 rpm for 5 min at 4 ℃. The serum will be immediately separated and stored at -70 ℃. Serum adiponectin will be assessed through enzyme-linked immunosorbent assay (ELISA) kits according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahim A. Sadek, Professor, Study Director — Sohag University; Abdelhady R. Abdel-Gawad, Lecturer, Study Chair — Sohag University; Elsayed M. Abdelkreem, Lecturer, Study Chair — Sohag University
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided